CLINICAL TRIAL: NCT02836405
Title: Investigations of Neuroplasticity Mechanisms in Autism Spectrum Disorders
Brief Title: TMS for the Investigation of Brain Plasticity in Autism Spectrum Disorders
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alexander Rotenberg, Associate Professor of Neurology, Boston Children's Hospital
Other Study IDs: 00014965; 1R01MH100186-01A1 (NIH)
Record Dates: First submitted 2016-05-13; First posted 2016-07-19 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability
Keywords: Autism; ASD; Autistic Disorder; Pervasive Development Disorders; Pervasive Child Development Disorders; Asperger's Syndrome; Transcranial Magnetic Stimulation; TMS; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability; Autistic Disorder; Child Development Disorders, Pervasive; Asperger Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva sample for genetic testing (optional)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Autism Spectrum Disorder (ASD): Individuals diagnosed with an Autism Spectrum Disorder (ASD) will receive transcranial magnetic stimulation (TMS) to measure brain plasticity.
  Interventions: Device: Transcranial Magnetic Stimulation
- Healthy Control: Typically developing individuals without a history of autism will receive transcranial magnetic stimulation (TMS) to measure brain plasticity.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Single pulses of TMS as well as continuous theta burst stimulation (cTBS) will be applied to the motor cortex.

SUMMARY:
The main purpose is to study brain plasticity (the changes that occur in the brain through experience) in individuals with autism spectrum disorder (ASD). Research suggests that during development, the brains of individuals with ASD may change in response to their experiences differently than the brains of typically developing individuals. Investigators want to understand why and how this difference may contribute to the symptoms of ASD.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are diagnosed clinically, based on key symptoms. As ASD phenotypic variability is large, and symptoms can manifest at different ages and degrees, the clinical diagnosis is challenging. To date, there remains an unmet need for a valid and reliable endophenotype that would facilitate ASD diagnosis early in life, enable efficient study of ASD risk factors, and eventually serve as a useful biomarker to inform the development of effective therapies and assess treatment response in future clinical trials.

As compared with behavioral or neuroimaging methods, transcranial magnetic stimulation (TMS) offers the advantage of providing behaviorally independent results that are largely unaffected by attention or cognitive ability. Therefore, a TMS based endophenotype may be applicable to all individuals across the autism spectrum.

At Boston Children's Hospital, each subject's participation in the study will consist of four visits: two screening visits, and two TMS sessions. At Beth Israel Deaconess Medical Center, each subject's participation will consist of three visits: one screening visit, and two TMS sessions. Each screening visit is expected to last between 2-3 hours, during which participants will first provide informed consent. Participants will then receive a thorough medical examination by a neurologist, and a neuropsychological evaluation (including IQ measures and ASD specific evaluations). If eligible to continue, participants will then come back for two identical TMS visits, that are spaced 1-5 weeks apart. These visits are expected to last between 3-4 hours, and include the TMS measures of brain plasticity.

ELIGIBILITY:
Inclusion Criteria at Boston Children's Hospital (children):

* For ASD group:

  1. Clinical diagnosis of a disorder on the autism spectrum.
  2. Assessment using the Autism Diagnostic Observation Schedule.
  3. Assessment using the Autism Diagnostic Interview-Revised.
  4. Children ages 6-16.
  5. IQ>70.
  6. Verbal.

Inclusion Criteria at Beth Israel Deaconess Medical Center (adults):

* For ASD group:

  1. Clinical diagnosis of a disorder on the autism spectrum.
  2. Assessment using the Autism Diagnostic Observation Schedule.
  3. Adults ages 21-65.

Exclusion Criteria:

* Intracranial pathology, cerebral palsy, history of severe head injury, significant dysmorphology, or known intracranial lesion.
* History of fainting spells of unknown or undetermined etiology.
* History of head injury resulting in prolonged loss of consciousness.
* History of seizures, diagnosis of epilepsy, or immediate family history of epilepsy.
* Any progressive neurological disorder or signs of intracranial pressure.
* Chronic uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure.
* Metal implants or devices.
* Substance abuse or dependence within the past six months.
* Certain prescription medications that decrease cortical seizure threshold.
* Pregnancy.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults diagnosed with an Autism Spectrum Disorder (ASD), as well as controls.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2015-05; Primary Completion 2020-04 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Percent of baseline TMS-induced measures of human synaptic plasticity | 120 minutes after cTBS
  Synaptic plasticity will be measured using the MEPs in response to cTBS. Baseline MEPs will be calculated before cTBS, and at different time points following cTBS up to 120 minutes. The investigators will compare post-cTBS MEPs to the baseline MEPs to calculate the percent change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rotenberg, MD, PhD, Principal Investigator — Boston Children's Hospital; Alvaro Pascual-Leone, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No